CLINICAL TRIAL: NCT00004236
Title: A Phase II Study of Caelyx in the Treatment of Advanced Gastric Cancer
Brief Title: Liposomal Doxorubicin in Treating Patients With Advanced Stomach Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067480; LRI-IND.02-3/98; EU-99034
Record Dates: First submitted 2000-01-28; First posted 2004-06-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2000-12

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating patients who have advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine overall survival, time to disease progression, objective reponse rate, safety profile, and quality of life in patients with inoperable gastric adenocarcinoma when treated with doxorubicin HCl liposome.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 1 hour every 4 weeks. Treatment continues for up to 6 courses in the absence of unacceptable toxicity or disease progression. Patients with responding disease may continue therapy past the 6 courses until documented disease progression. Quality of life is assessed prior to every treatment course. All patients are followed at 1 month. Patients with stable or responding disease are then followed every 3 months until death.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced gastric adenocarcinoma, including adenocarcinoma of the esophagogastric junction Evaluable disease No CNS involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin normal AST or ALT less than 3 times upper limit of normal (ULN) (5 times ULN if documented liver metastases) Renal: Creatinine less than 1.5 times ULN Cardiovascular: LVEF normal No history of New York Heart Association class II-IV heart disease with congestive heart failure No unstable cardiovascular disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other prior primary cancer within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix No hypersensitivity to anthracycline therapy No history of severe hypersensitivity reactions to products containing Chremophor EL (e.g., cyclosporine or teniposide for injection concentrate) No other significant medical disorder (e.g., active uncontrolled infection) that would preclude study treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior chemotherapy for metastatic disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to less than 1/3 of hematopoietic sites and recovered Surgery: Not specified Other: At least 30 days since other prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth O'Byrne, MD, Study Chair — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, England, United Kingdom